CLINICAL TRIAL: NCT01507571
Title: Implementation and Evaluation of Dignity Therapy in Denmark
Acronym: DignityDK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Mogens Groenvold, MD, PhD, D.M.Sci., Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DignityTherapyDK 01; PP04011 (Other Grant/Funding Number: Danish Cancer Society)
Record Dates: First submitted 2011-11-11; First posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Cancer
Keywords: Incurable cancer; Palliative care; Dignity Therapy; Loss of dignity; Patient Dignity Intventory; Eortc QLQ-C15-PAL; Structured Interview for Symptoms and Concerns; Hospital Anxiety and Depression Scale
MeSH Terms: conditions — Neoplasms; Depression | interventions — Dignity Therapy; Psychosocial Intervention; Terminal Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dignity Therapy (Experimental)
  Interventions: Other: Dignity Therapy

INTERVENTIONS:
Other: Dignity Therapy — Dignity Therapy is a brief psychotherapeutic intervention consisting of:
  1. a tape-recorded session with the patient using the DT question protocol
  2. Transcription of the interview, which is then edited
  3. A session where the edited transcript is returned to the patient who can give it to family members or friends.
  If needed, one or more sessions are added. Dt allows the patient to give voice to the matters of importance concerning himself and his loved ones. Its purpose is to enhance sense of meaning, purpose and worth. It also gives the opportunity to leave something behind to be remembered by.
  Other Names: Psychotherapeutic intervention; Psychosocial intervention; End of life care

SUMMARY:
The purpose of the study is to investigate whether Danish patients with incurable cancer have a need of, interest in and benefit from Dignity Therapy.

DETAILED DESCRIPTION:
Research in palliative care has primarily focused on physical and psychological symptoms. Research in other psychosocial and existential problems has been sparse. Loss of dignity as a consequence of serious illness may be an important cause of suffering. The research team of the Canadian psychiatrist and professor, Harvey Chochinov has investigated the concept of dignity and developed the psychosocial intervention 'Dignity Therapy' (DT). The preliminary research results were promising.

Research questions: Do Danish cancer patients have a need of, interest in, and benefit from DT? Methods: DT consists of an interview revolving around the patient's life, values, and accomplishments and is also an opportunity to leave messages and words of hope and compassion for friends and family. The interview is audio taped, transcribed, and edited together with the patient, and made into a tangible document, which the patient can give to his/her relatives. The project consists of three parts: (1) a cross-sectional investigation of the prevalence of loss of dignity and related symptoms/problems among at least 200 incurable cancer patients. (2) A feasibility study, testing the intervention in terms of relevance and the need of any modifications in relation to Danish patients. (3) An evaluation study testing the effect of and satisfaction with DT.

At least 80 patients are planned for the feasibility and evaluation studies. Questionnaires are used for detection of loss of dignity and as measures of effect. These will be administered before the intervention and, along with a semi-structured evaluation questionnaire, right after the intervention, when the document is received and again approximately two weeks later.

The duration of the intervention (DT) varies markedly between patients. In some cases the process (interview, transcription, editing of document, and the final meeting where the document is given back to the patient) is completed urgently in a few days, whereas in other cases, the patient prefers a slower pace, and may want to sub-divide the interview into two or more parts. Also, when presented with the document, some patients want to have something changed or they want add material. This variation is seen as intentional, as it illustrates that the process is tailored to the patient's wishes.

As stated, the effect of the DT intervention is evaluated at completion of the intervention, i.e. when the final document is given back to the patient, and about two weeks later. Due to process described above, the time from the first measurement (before intervention) to the second measurement (which takes places at completion of the intervention) therefore varies considerably (median 36 days after baseline, range 7-121 days).

Perspective: If Danish patients have a need of, an interest in and benefit from DT, it can be offered to Danish patients admitted to palliative care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of incurable cancer,
* 18 years or older,
* informed of diagnosis and the incurable prognosis.

Exclusion Criteria:

* dementia and other cognitive impairment,
* physical limitations,
* sufficient to preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Sense of dignity | Pre-post intervention (when the document was recieved by the patient), and again two weeks later.
  Measured with the Structured Interview for Symptoms and Concerns (SISC)

SECONDARY OUTCOMES:
Hopelessness | Pre-post intervention (when the document was recieved by the patient), and again two weeks later.
  Measured with the Structured Interview for Symptoms and Concerns (SISC)
Anxiety | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Hospital anxiety and depression scale
Depression | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Hospital Anxiety and Depression scale
Not able to perform tasks of daily living | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Patient Dignity Inventory
Suffering | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured with the Structured Interview for Symptoms and Concerns
performance status | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Palliative Performance Scale v2
Communication | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Structured Interview for Symptoms and Concerns
Social Contact | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the Structured Interview for Symptoms and Concerns
Depression | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured with the Structured Interview for Symptoms and Concerns
Not able to attend to bodily functions | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Physically distressing symptoms | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling how I look has changed | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling depressed | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling anxious | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling uncertain | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Worried about future | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not able to think clearly | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not able to continue usual routines | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling no longer who I was | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not feeling worthwhile or valued | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not able to carry out important roles | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling life no longer has meaning or purpose | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling of not having made a meaningful contribution | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling of unfinished business | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Concerns regarding spiritual life | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling like a burden to others | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling of not having control | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Feeling of reduced privacy | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not feeling supported by friends or family | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not feeling supported by health care providers | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not feeling able to mentally fight illness | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not being able to accept things as they are | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Not being treated with respect | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Item from the Patient Dignity Inventory
Physical function | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Emotional function | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Overall quality of life | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Fatigue | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Nausea / Vomiting | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Pain | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Dyspnoea | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Insomnia | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Appetite loss | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL
Constipation | Pre-post intervention (when the document was received by the patient), and again two weeks later.
  Measured on the EORTC QLQ-C15-PAL

CONTACTS AND LOCATIONS:
Overall Officials: Mogens Groenvold, MD PhD DSci, Principal Investigator — Bispebjerg Hospital/ Department of Public Health, Faculty of Health Sciences, University of Copenhagen
Locations (2):
- Denmark (2):
  - Department of Palliative Medicine, Copenhagen
  - Sankt Lukas Hospice, Hellerup

REFERENCES:
- [Result] Houmann LJ, Rydahl-Hansen S, Chochinov HM, Kristjanson LJ, Groenvold M. Testing the feasibility of the Dignity Therapy interview: adaptation for the Danish culture. BMC Palliat Care. 2010 Sep 22;9:21. doi: 10.1186/1472-684X-9-21. PMID 20860786
- [Derived] Houmann LJ, Chochinov HM, Kristjanson LJ, Petersen MA, Groenvold M. A prospective evaluation of Dignity Therapy in advanced cancer patients admitted to palliative care. Palliat Med. 2014 May;28(5):448-58. doi: 10.1177/0269216313514883. Epub 2013 Dec 5. PMID 24311296